CLINICAL TRIAL: NCT03467100
Title: Phase 1, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Oral Doses of XEN901 in Healthy Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Oral Doses of XEN901
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XPF-006-101; 2017-004046-26 (EudraCT Number); QCL118145 (Other: Quotient Sciences Study Number)
Record Dates: First submitted 2018-03-02; First posted 2018-03-15 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XEN901 (Experimental): Single ascending dose: Single oral dose for each cohort; Multiple ascending dose: 7 days of single oral dose twice daily for each cohort
  Interventions: Drug: XEN901
- Placebo (Placebo Comparator): Single Ascending Dose: Single oral dose for each cohort; Multiple Ascending Dose: 7 days of single oral dose twice daily for each cohort
  Interventions: Drug: Inert Ingredients Oral Product

INTERVENTIONS:
Drug: XEN901 — Capsule filled with XEN901
  Arms: XEN901
Drug: Inert Ingredients Oral Product — Placebo capsule
  Arms: Placebo

SUMMARY:
The XEN901 Phase 1 clinical trial is a randomized, double-blind, placebo-controlled study that will evaluate the safety, tolerability and pharmacokinetics (PK) of both single ascending doses (SAD) and multiple ascending doses (MAD) of XEN901 in healthy subjects. It is estimated there will be approximately 64 subjects in the planned SAD and MAD cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male or females aged between 18 and 55 years inclusive with a body mass index (BMI) between 18.5 and 32.0 kg/m2
* Must agree to use effective methods of contraception, if applicable
* Able to swallow capsules
* Able to provide written, personally signed and dated Informed Consent Form

Key Exclusion Criteria:

* Any history of seizures
* Any current and relevant history of significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk, affect clinical or laboratory results, or the subject's ability to participate in the study
* Answering "yes" to any of the questions within the Columbia Suicide Severity Rating Scale
* Mental incapacity or language barriers precluding adequate understanding, cooperation, and compliance with the study
* No prescription or over-the-counter (OTC) medications (except hormonal contraception), herbal or dietary supplements OTC medications 14 days prior to dosing to study end
* No smoking 60 days prior to dosing to study end
* Any clinically significant abnormalities in vital signs, ECG, physical exam, or laboratory evaluations

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as assessed by CTCAE v4.03 | From screening (28 days prior to Day 1) through to 30 days post-final dose
  To assess AEs as a criteria of safety and tolerability
Resting 12-lead electrocardiogram (ECG) | At screening (28 days prior to Day 1) through to 7 days post-final dose
  To assess 12-lead ECG intervals (PR, QRS, QTcF, RR) as a criteria of safety and tolerability
Number of participants with vital sign abnormalities | At screening (28 days prior to Day 1) through to 7 days post-final dose
  To assess vital signs as a criteria of safety and tolerability

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day 1 predose through to 7 days post-final dose
  Cmax is the maximum observed plasma concentration in ng/mL
Time to the Maximum Observed Plasma Concentration (Tmax) | Day 1 predose through to 7 days post-final dose
  Tmax is the time in hours to reach Cmax following dosing
Terminal elimination half-life (t1/2) | Day 1 predose through to 7 days post-final dose
  The time in hours required for the plasma level of the study drug to decrease by one-half during the terminal elimination phase
Area Under the Plasma Concentration-Time Curve from Time Zero to the Time of the Last Quantifiable Plasma Concentration (AUC0-last) | Day 1 predose through to 7 days post-final dose
  The area under the plasma concentration-time curve [in ng.h/mL] from time zero to the time corresponding to the last quantifiable plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Beatch, PhD, Study Director — Xenon Pharmaceuticals Inc.
Locations (1):
- Quotient Sciences, Ruddington, United Kingdom